CLINICAL TRIAL: NCT06809166
Title: Identifying the Short-Term Neurobiological, Metabolic and Behavioural Effects of CONTRAVE as Potential Mechanisms of Weight Loss in Adults With Obesity: A Randomized, Double-Blind, Placebo-Controlled Pilot Trial
Brief Title: Metabolic and Behavioural Effects of CONTRAVE as Potential Mechanisms of Weight Loss in Adults With Obesity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Royal's Institute of Mental Health Research (Other)
Collaborators: University of Ottawa (Other); The Royal Ottawa Mental Health Centre (Other); Bausch Health, Canada Inc. (Unknown); Cheo Research Institute (Other); LEAF Weight Management Clinic (Unknown)
Responsible Party: Principal Investigator, Dr. Natalia Jaworska, Director, The Royal's Institute of Mental Health Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023004
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Weight Loss; Weight Management; Dietary Intervention; Obesity/Therapy
Keywords: contrave; EEG; MRI; weight loss; appetitive behaviour; executive functioning; mood and weight loss; mood; body composition; symptoms of anxiety; symptoms of depression; energy expenditure; appetite; energy intake; food reward; reward processing; motivation; effort expenditure; delay discounting; brain activation; event related potentials; brain electrical activity
MeSH Terms: conditions — Obesity; Weight Loss; Depression | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination; Naltrexone; Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTRAVE (Experimental): A diet program + CONTRAVE®
  Interventions: Drug: Contrave; Behavioral: Diet Program
- Placebo (Placebo Comparator): Diet Program + Placebo
  Interventions: Drug: Placebo; Behavioral: Diet Program

INTERVENTIONS:
Drug: Contrave — CONTRAVE® will be titrated up to a therapeutic dose (Naltrexone 32mg/Bupropion 360mg) over a 4-week period as per clinical guidelines, and what is typical in the LEAF clinic. Dose recommendation for CONTRAVE® is tablet based, with each tablet containing 8mg of naltrexone and 90mg of bupropion. The maximum recommended daily dose is two tablets, administered orally, twice daily (32mg/360mg), taken once in the morning and once in the evening. Tablets and dispensing schedule will be done under the oversight of The Royal pharmacy (i.e., they will instruct the participants on the dosing schedule).
  Medication adherence and side effects will be reported daily using our online data capture system (REDCap) (approximately 1min) starting on the evening of the first dose of administration. If adverse events are significantly concerning, there is a mechanism in place for dealing with such events.
  Other Names: Naltrexone/Bupropion-NB
  Arms: CONTRAVE
Drug: Placebo — Placebo intervention will follow the exact same protocol in terms of tablet numbers as the CONTRAVE intervention.
  Generic Placebo pills will be packaged by The Royal Pharmacy into blister packs identical to Contrave.
  Other Names: Vitamin Pill
  Arms: Placebo
Behavioral: Diet Program — All participants will receive an individualized dietary intervention with appropriate energy restriction from registered dietitians at Dr. Shiau's LEAF weight management clinic (called the 4-week BUDS program, which is offered to clients with obesity at the LEAF clinic). The program involves weekly touch points with a registered dietitian, and meal planning/coaching and integrates a partial meal replacement with a commercial shake.

SUMMARY:
Obesity is a common chronic disease linked with increased risk for other illnesses and earlier death. Our team and others have shown that many bodily and psychological changes occur when individuals are on calorie-restricted diets. These changes might undermine dietary adherence and help to explain the relatively poor long-term efficacy of diets. These include increased appetite, increased food 'value' and 'wanting' that leads to overconsumption. Other factors include more sensitive sensory cues (e.g., smelling), higher food liking and craving, and a drop in resting energy expenditure (REE). REE has been shown to predict weight regain.

The standard care for obesity may include the use of the weight-loss drug CONTRAVE®. The Federal Drug Agency (FDA) and Health Canada have approved this drug for weight management and obesity treatment.

Although CONTRAVE® was designed to reduce appetite, food-related impulsivity and cravings, its mechanisms of action are unclear. In other words, the effects of CONTRAVE® on REE, executive function, and brain changes remain unknown in humans. A better understanding of how this drug works on the brain and body could lead to improvements in obesity management in the future.

As such, the goal of this research is to study the effects of 4 weeks of CONTRAVE® (+ diet program) vs. control (placebo pill + diet program) on mood, body composition changes, biological/metabolic measures, and brain measures.

Adults aged 18-64 with obesity will be randomized to one of two groups: diet + CONTRAVE® (CONTRAVE®, 20 participants) or diet + Placebo (Placebo, 20 participants). Both groups will be assigned the same study procedures for the entire study duration. The only difference is that Group 1 will receive CONTRAVE® while Group 2 will receive a placebo (non-medical) pill.

The study design and intervention is as follows:

Participants who meet all the telephone screening criteria will be invited to the Clinical EEG & Neuroimaging Laboratory at The Royal's IMHR for an in-person screening and test-dose session. Participants who are cleared by the study physician, Dr. Pierre Blier, during the in-person screening will be enrolled in the 4-weeks trial.

After the in-person screening visit, participants will attend two baseline testing visits (before starting the medication + diet program). The first will occur at the Behavioural and Metabolic Research Unit at the University of Ottawa. During this in-person visit, measures of body composition, resting energy expenditure, appetite, food craving, impulsivity, eating behaviours, taste and odour sensitivity, energy intake, and food preference will be collected.

The second baseline visit (within a week of the first one) will occur at The Royal/IMHR. During this visit, participants will be asked to complete questionnaires. They will undergo an EEG recording while resting and performing computer tasks. They will also get a brain imaging scan, during which they are asked to rest and complete a computer task.

Both testing sessions (University of Ottawa and Royal Ottawa testing sessions) will be repeated after four weeks of treatment. The section below provides further description and timing of these visits.

As part of the treatment, you will receive an individualized dietary intervention with appropriate energy restriction from a registered dietitian at Dr. Judy Shiau's LEAF weight management clinic (called the 4-week BUDS program). The program involves weekly touch points with a registered dietitian and meal planning/coaching. The diet intervention will commence the same week as the start of the placebo/CONTRAVE®.

During the 4-week intervention, participants will be asked to complete online questionnaires at various times.

DETAILED DESCRIPTION:
Detailed Description

This study is a two-arm, randomized, double-blind, placebo-controlled design, wherein N=40 adults aged 18-64 years with obesity (body mass index [BMI] > 30) and who meet all inclusion criteria (outlined below) will be randomized to one of two groups: Diet + CONTRAVE® (CONTRAVE®, N=20) or diet + Placebo (Placebo, N=20).

Participants will be randomized 1:1 per condition using a randomization program (computer-program). Each participant will be assigned a unique identifier code. Master codes containing the link between the identification code and name of the individual will be stored on a password-protected master file (excel) that will be saved on hospital servers (password-protected) in the Clinical EEG & Neuroimaging Laboratory (Co-PI: N. Jaworska). All hard-copies of confidential information (e.g., screening documents, consent forms) will be housed in secured cabinets within the Clinical EEG Laboratory.

Recruitment for this study will occur from Dr. J. Shiau's LEAF Weight Management Clinic. Following initial assessment of needs, a staff member of the LEAF clinic will mention this study and ask interested individuals to complete an online form as initial registration in the study. These potential participants will be contacted by research staff who are not affiliated with the LEAF clinic (i.e., research assistant or trainees who are part of the research team); the research personnel will then phone interested participants to explain the study and associated risks and benefits of participating. Participants who do not wish to participate in the research study after details are provided, will continue with the normal intake process at the LEAF clinic. Participants who wish to participate will complete a telephone screening questionnaire with the research staff. Eligible participants will be booked for an in-person screening session at The Royal Ottawa Mental Health Centre.

Screening and Testing Sessions Overview:

Participants will have 5 in-person laboratory visits (Clinical EEG & Neuroimaging Laboratory, under the direction of Dr. Natalia Jaworska, at The Royal/IMHR; and, Behavioural and Metabolic Research Laboratory, under the direction of Dr. Eric Doucet, at the University of Ottawa). Specifically,

* Visit 1: in-person screening and test dose visit at the Clinical EEG & Neuroimaging Lab, at The Royal;
* Visit 2: baseline metabolics/cognition/food craving assessment at the Behavioural and Metabolic Research Laboratory, University of Ottawa;
* Visit 3: baseline EEG/MRI imaging at the Clinical EEG and Neuroimaging Laboratory at The Royal;
* Visit 4: 4-week post-intervention metabolics/cognition/food craving assessment at the Behavioural and Metabolic Research Laboratory, University of Ottawa;
* Visit 5: 4-week post-intervention EEG/MRI imaging at the Clinical EEG and Neuroimaging Laboratory at The Royal.

Phone Screening:

Participants will be recruited from the LEAF clinic. Those who are interested in participating complete an online registration form. They will then be contacted by research study personnel and screened over the phone, regarding basic inclusion criteria. The study will also be explained. Following successful phone screening, an in-person screening visit and test dose (administered by The Royal pharmacy and overseen by Dr. Pierre Blier) visit will be scheduled at the IMHR (Dr. Jaworska's laboratory). Only participants who have been cleared medically by the LEAF clinic/Dr. Judy Shiau will be referred to this study.

In Person Screening:

This will occur at The Royal. The informed consent will be carried out, and any questions will be addressed and documented directly on the consent form. Second, a brief clinical assessment (to ensure that outstanding inclusion and exclusion criteria are met), using modules from the MINI (Mini International Neuropsychological Inventory) including the mood module, substance use module, psychotic disorders module, and eating disorders module (approximately 30min). Heart rate and blood pressure will then be measured reviewed by Dr. Pierre Blier.

Test Dose Administration (as part of In Person Screening Session):

Subsequently (during the in-person screening), The Royal's pharmacy would issue one test dose of the drug placebo or CONTRAVE® based on the participant drug randomization. This pill would be given to the participant. The test dose will be 1 tablet of placebo or CONTAVE® (8mg Naltrex/90 mg Buproprion). The participant and study doctor and research staff will be blind to treatment (they will not know whether they will be given CONTRAVE® or placebo). Only research personnel from the laboratory -not directly related to this study- and the pharmacy team will know what the randomization is (i.e., what participant is receiving what drug). The participant would take the pill along with crackers/light snack in Dr. Blier's laboratory (as CONTRAVE® should be taken with food) and watch a movie and/or read a book or work (participant preference) for 3 hours in one of the examination chambers in the Mood Disorders Unit.

After 3 hours of ingesting the test dose, and -at that time- exhibiting no/minimal adverse symptoms (i.e., most common adverse events symptoms include nausea, vomiting, constipation, stomach pain, headache, dizziness, trouble sleeping, increased sweating, flushing, and dry mouth or strange taste in the mouth), participants will be free to go home. If any concerning, unexpected or severe adverse events linger, the clinician will be responsible for managing the participant, in accordance with standard medical procedures (Dr. Blier).

Based on tolerability to the test dose, in consultation with the participant and the clinician, the participant will be invited to continue (or not) with the remainder of the study. A week after the test dose, eligible participants (i.e., those who tolerate the test dose, and wish to proceed) will be booked for their baseline session. Those participants who are deemed to be intolerant to the test-dose will be counted screen failures.

Body measures (e.g., weight, height, approximately 5min) will be collected and the neurocognitive battery (NIH Toolbox; approximately 30min); The neurocognitive battery, which assesses various cognitive domains (e.g., spatial memory, verbal memory, attention, inhibition) will be used to characterize the sample, and explore whether CONTRAVE® changes cognitive profiles. Participants will also undergo a session in the mock scanner situated at the BIC to ensure that they can fit into the bore of the magnet and are comfortable with neuroimaging (approximately 15min). For participants who are not comfortable with scanning/cannot fit into the scanner, they will be invited to participate in all the other elements of the proposed work (outlined below), apart from the neuroimaging.

Baseline Session (uOttawa):

Participants will complete a baseline assessment in the Behavioural and Metabolic Research Laboratory, University of Ottawa under Dr. Doucet's supervision. In his laboratory, they measure the following:

* Body Composition
* Resting and Post-Prandial Energy Expenditure
* Food palatability and appetite ratings
* Food Craving
* Food Reinforcement
* Changes in eating behavior traits/styles (Restrained, Emotional and External eating)
* Taste sensitivity/olfaction to a variety of flavors (e.g., sweet, salty, bitter etc)
* Lunch will be served and participants will be asked to self-select foods from a food menu. They will be instructed to eat as much as they desire of these foods. Energy intake and food preferences will then be assessed from the weight of the different foods consumed.

Baseline Session (The Royal):

The baseline session will take place in the Clinical EEG & Neuroimaging Lab under the supervision of Dr. Jaworska. The following measures will be collected:

A) Electroencephalographic (EEG) & Autonomic Nervous System (ANS) assessments:

EEG & ANS assessments involve using a 64 or 32-channel EEG system along with additional electrodes for ANS indices like HRV and SCR. Setup by experienced personnel takes 20-30min. Data collection includes:

* 5-min eyes closed EEG and ANS recordings for baseline neural features.
* EEG and ERPs during a food impulsivity task, evaluating impulsivity for various food and non-food stimuli.
* A reward task assessing effort for rewards, with specific ERPs reflecting reward and error processing.
* Measurement of HRV and SCR during each task.

B) Neuroimaging:

Participants qualifying for neuroimaging will undergo a 30min brain scan at the Brain Imaging Centre using a 3T PET-MR Siemen's scanner.

Scans include:

* Resting-state fMRI focusing on connectivity and activity in appetitive, reward, and cognitive regions.
* Task-based fMRI comparing responses to high-caloric vs. low-caloric vs. neutral images
* High-resolution structural imaging (MEMPRAGE) to assess anatomical features in obesity, compared with healthy-weight data.
* If time permits, magnetic resonance spectroscopy (MRS) to assess neurochemical composition in the ventral striatum/nucleus accumbens, primarily related to reward processing.

C) Clinical measures include self-report depression and anxiety questionnaires.

D) Sleep and activity data will be collected via daily logs and accelerometry.

Intervention:

Following the completion of the baseline sessions (TheRoyal/uOttawa), participants will begin their interventions, which will include starting their medication (placebo or CONTRAVE®, based on randomization) and LEAF diet program. Participants will obtain their 4-week prescriptions from The Royal pharmacy after their in-person screening visit at The Royal. However, they will be told not to commence their treatment until they complete both baseline testing sessions and are instructed to start the medication (i.e., start of intervention week 1). The prescription for the CONTRAVE® and placebo will be filled out by the responsible physician, Dr. Judy Shiau; this will be faxed/send directly to the The Royals' pharmacy prior to the participants' arrival for their in-person screening visit.

The diet intervention will commence the same day as the start of the placebo/CONTRAVE® administration. Diet adherence and food intake will be measured daily using our online data capture system (REDCap) (approximately 1min) (carried out the same time as the sleep and adverse events questionnaire). Food journaling will be carried out through the Eat.Love platform as part of the diet coaching that will be guided by the LEAF clinic.

Monitoring:

Daily monitoring of side effects/adverse events will be conducted by a devoted research team member in Dr. Jaworska's laboratory using our REDCap during the first week of use, and weekly thereafter (i.e., mid of week 2, week 3 and week 4). A copy of all adverse events ratings for all active participants will be shared with Dr. Shiau on a weekly basis for clinical review and assessment, which Dr. Shiau will then sign, date and return to the research team. If participants experience moderate adverse events, the research personnel will inform Dr. Shiau immediately, and she can recommend dose adjustments. Participants who experience unexpected/severe adverse events will be instructed to contact the LEAF clinic to report this immediately (as per LEAF protocols). Severe adverse events will be handled as per regulated standards of care. If Dr. Shiau (responsible physician) deems that the adverse events are severe, she might advise the participant to discontinue the drug. This will be communicated to the research team (a member of the research team will thus break the blind to determine whether the drug was placebo or CONTRAVE®). Discontinuation due to adverse symptoms will be documented in the participant file.

Post-Intervention Assessment:

Following the completion of the 4-weeks of medication and diet program, participants will complete the exact same testing sessions as during the baseline sessions. The sessions will be carried out as close as possible to the end of the 4-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are able to provide written informed consent prior to the initiation of any protocol-required procedures
2. Have been referred to the LEAF clinic by their physician or have self-referred to the LEAF clinic for weight loss, and have been deemed appropriate for weight loss treatment offered by the LEAF clinic (i.e., these criteria are at the discretion of the clinical team at the LEAF clinic, outlined below in the exclusion criteria section).
3. Adults: aged 18-64 years of age (gender and sex will be noted; recruitment is all-gender inclusive).
4. Have a BMI>30.
5. Have normal or corrected vision as some of the study aspects will involve viewing/responding to visual stimuli.
6. Understand and speak English (as instructions for study criteria will be provided in English).
7. Able to participate in the study protocol as described, e.g. have a means of getting to the laboratories and no major mobility issues to the extent that protocols cannot be followed (details below).
8. Access to a secure internet connection (for virtual appointments with members of the LEAF clinic).

Exclusion Criteria:

1. Reporting severe depression or reporting significant suicidal ideation, or history of bipolar disorder or psychosis (i.e., major psychiatric condition; this will be ascertained during the screening carried out by research personnel, in keeping with our standard protocols in Dr. Jaworska's laboratory).***
2. Current use of antidepressants, thyroid medication, or any medication that could affect appetite, or seizure threshold (e.g.., bupropion, tamoxifen, thioridazine).
3. Uncontrolled hypertension.
4. History of cardiac defects or symptoms suggestive of any cardiac condition (not including coronary artery disease).
5. Presence of diabetes.
6. Current or past history of addictions or substance use disorder, including undergoing abrupt discontinuation of alcohol, benzodiazepines, barbiturates, and antiepileptic drugs.
7. History of eating disorder (including Binge Eating Disorder, Bulimia Nervosa or Anorexia Nervosa).
8. History of glaucoma.
9. Personal or family history of seizure disorders.
10. Currently taking MAO inhibitors (within 14 days), pressor agents, coumadin, anticonvulsants, or phenylbutazone, or other bupropion-containing products (such as Wellbutrin, Wellbutrin SR, Wellbutrin XL, Aplenzin or Zyban), or CYP2B6 inhibitors (e.g. ticlopidine or clopidogrel).
11. History of thyroid disease, chronic liver, or renal disease.
12. Chronic use of opioid, opiate agonist (Methadone) or partial agonists (Buprenorphine).
13. Currently pregnant or planning to become pregnant during the intervention or currently nursing. Pregnancy urine test will be conducted during the in-person screening session in the laboratory.***
14. No known allergy to any of the ingredients in CONTRAVE® (e.g. lactose).
15. Hereditary problems of galactose intolerance, lactase deficiency or glucose-galactose malabsorption.
16. Current use of obesity medications such as liraglutide or semaglutide or orlistat.
17. Current use of medication indicated in patient living with ADHD (e.g., Vivanse/Concerta) which are known to have metabolic impacts.

    There are several additional exclusionary criteria, established by research personnel in Dr. Jaworska's laboratory (i.e., not part of LEAF intake) that preclude participation in the brain imaging/magnetic resonance imaging (MRI) and EEG, these include:
18. Severe claustrophobia.
19. Inability to lie still in the scanner for approximately 30min.
20. Metal in the body that cannot be removed and might pose a safety risk to the participant.
21. History of concussion (loss of consciousness for >5-min).
22. Major neurological illness, such as, epilepsy, stroke, tumours (as this would interfere with the interpretation of the MRI data).
23. Obesity to the extent that the participant cannot fit into the scanner. This will be established by ensuring that the individual can fit into the mock scanner at the Brain Imaging Centre (BIC) of The Royal. If a person cannot fit into the mock scanner, it is unlikely that the person can fit into the real scanner.
24. Testing positive for illicit drugs and cannabis (this will be established using a drug test that will be administered in the Clinical EEG & Neuroimaging laboratory at the Institute of Mental Health Research [IMHR]). Participants who are cannabis users will be invited to participate in the study so long as they can abstain from cannabis use for approximately 2weeks prior to the baseline session and approximately 2weeks before final assessment. Ideally, participants would also abstain from cannabis use during treatment, but, this will not be tested/enforced.
25. Ability to abstain from nicotine/tobacco and caffeine for 3h prior to the baseline testing/EEG recordings, as both substances influence EEG activity.

    NOTE: If a participant cannot participate in the MRI aspect of the study (i.e., due to the above exclusion criteria), they will still be able to participate in the research study (apart from the MRI component). All MRI/EEG exclusion criteria will be established during the screening/clinical interview carried out by trained research staff from Dr. Jaworska's laboratory (details below).

    One final exclusion criterion is as follows:
26. Unable to tolerate the test dose of CONTRAVE® (details below). Such individuals would not participate in further elements of the research, but, would continue with their treatment through the LEAF clinic (as determined by the LEAF clinic, per their clinical management program).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
MRI Modalities | 4 weeks
  Four MRI modalities will be collected during two identical 45-minute MRI session: one at baseline and another 4-weeks post placebo or Contrave. The first modality is an 8-minute resting-state functional MRI to assess brain activity at rest. Second is a 7-minute structural scan, which will allow us to explore potential changes in brain volume. Third, is a 12-minute task-based functional MRI scan where participants are presented with images of food/non-food visual cues, allowing us to assess brain activity in response to different cues. Last is a 9-minute neuromelanin scan, which allows us to visualize neuromelanin in the brain. Neuromelanin is present in brain regions implicated in the brain's reward system and is a marker of dopamine, which is highly involved in motivation and reward. This exploratory scan will help elude neuromelanin levels and locus coeruleus contrast in individuals with obesity and whether there are correlations with other neuroimaging/clinical measures.
Changes in body weight/composition | 4 weeks
  Dual Energy X-ray Absorptiometry (DEXA) will be used to measure lean mass, fat mass and percent body fat (Lunar Prodigy, GE Medical Systems)
Brain Activity EEG at Rest | 4 weeks (pre and post contrave or placebo)
  Electroencephalography (EEG) at baseline and 4-weeks post placebo or Contrave.
  EEG will involve a 16-channel EEG system. Data collection includes resting EEG spectral power extracted from resting EEG and may include the following frequency bands:
  * Delta (1-4 Hz)
  * Theta (4-8 Hz)
  * Alpha (8-13 Hz)
  * Beta (13-30 Hz)
  * Gamma (>30 Hz)
  Analysis: Power is typically analyzed for each frequency band.
Brain Activity During Food Impulsivity Task | 4-weeks (pre and post contrave or placebo)
  EEG-derived event-related potentials (ERPs) will be assessed during a food impulsivity task (Go/No-Go task).
  Specifically, N2 and P3 ERP amplitudes (µV) and latencies (ms) will be measured in response to neutral objects trial, high calorie foods and low calorie foods trials.
  Behavioural measures, including correct and incorrect responses (%) and reaction times (%) will be measured as secondary outcome measures.
Brain Activity During EEFRT Task | 4-week (pre and post contrave or placebo)
  Using the Effort Expenditure for Rewards Task (EEfRT) specific ERPs associated with reward and error processing will be obtained.
  Specifically, ERP amplitudes (µV) and latencies (ms) for the Stimulus Preceding Negativity (SPN), and the P3 for the easy and hard trials will be analyzed separately.
  The number of times participants chose the easy vs. hard trials (difficulty) is analyzed as a measure of motivation.

SECONDARY OUTCOMES:
Hedonic Mechanisms | 4 weeks
  Food palatability and appetite ratings (hunger, fullness, desire to eat, and prospective food consumption) will be measured using a 100-mm Visual analog scale (VAS) at fasting, at 0, 30, 60, 90, 120, 180 min after a standardized breakfast administered in the laboratory. Changes in both state and trait-related food craving will be assessed by the self-reported Food Craving Questionnaire. The relative reinforcing value of snack foods in relation to healthy food alternatives will also be assessed.
  Lunch will be served at approximately 12h30. Participants will be asked to self-select foods from a food menu. They will be instructed to eat as much as they desire of these foods. Energy intake and food preferences will then be assessed from the weight of the different foods consumed.
Mood | 4 weeks
  Self-reports of depression and anxiety symptoms will be assessed using the Beck Depression Inventory (BDI) and the Generalized Anxiety Disorder (GAD-7).
  These will be collected on an iPad or pen-and-paper (as per participant's preference). Data collected on an iPad will be collected using REDCap (a data collection platform used/available at The Royal, which is known to comply with privacy standards; all imputed data will be only liked with the participant code).
  The active drug condition (contrave) may influence mood; thus, we will track mood changes before vs. after 4-weeks of intervention.
  Mood scores (i.e., anxiety and depression) will be used as covariates in the analyses of behavioural and brain activity (MRI, EEG, ERP) measures listed in the primary and secondary outcomes.
Metabolic Effects | 4 weeks
  Resting and Post-Prandial Energy Expenditure:
  Energy expenditure (EE) will be measured fasting and after a standardized breakfast with indirect calorimetry (Vmax Encore 29N metabolic cart by SensorMedics, Yorba Linda, CA, USA). (approximately 45 min for resting and then 30 min every hour for 2 hours after a standardized breakfast, which will be provided in the laboratory).
Executive Functioning | 4 weeks
  Measured with NIH cognition toolbox.
Behavioural and EEG During a Delay Discounting Task | 4 weeks (pre and post contrave or placebo)
  During a monetary delay discounting task, behavioural data will be collected and will include the number of times participants chose immediate vs delayed reward. Discount rate will also be examined.
  Spectral power derived from EEG data may be analyzed as a secondary measure.
Motivation Measures | 4 week
  Contrave may influence motivation; thus, we will track motivation changes before vs. after 4-weeks of intervention with the placebo and CONTRAVE®. Using the Behavioural Inhibition System (BIS) and Behavioural Activation System (BAS) will assess motivation and personality-related behaviours.
  These measures of motivation will be assessed in correlation with measures of:
  * eating, hunger and food craving collected with the Food Craving Questionnaire.
  * EEG and ERP measures collected during the food impulsivity task, the effort expenditure task, and the delay discounting task.
Autonomic Nervous System Measures | 4 weeks
  Using a BIOPAC and 5 electrodes, measures of heart rate variability and skin conductance will be collected during the EEG resting state, the food impulsivity task, the effort expenditure task, and the delay discounting task.
  Heart rate variability and skin conductance measures will be correlated with amplitude (µv), latency (ms), and behavioural (correct responses, incorrect responses, reaction times, number of hard vs easy trials, and immediate vs delayed reward measures extracted from the previously described tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blier, M.D., Ph.D, Principal Investigator — University of Ottawa
Locations (3):
- Canada (3):
  - LEAF Weight Managment Clinic, Ottawa, Ontario
  - Behavioural and Metabolic Research Unit, Ottawa, Ontario
  - University of Ottawa Institute of Mental Health Research, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No